CLINICAL TRIAL: NCT06820229
Title: 5-Fluorouracil Cream Versus Modified Carnoy's Solution As Adjunctive Methods In Treatment Of Odontogenic Keratocyst
Brief Title: Adjunctive Methods In Treatment Of Odontogenic Keratocyst
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohamed Kamal Eid Allam, Associate professor, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Research Ethics CommiOS07-22/2
Record Dates: First submitted 2025-02-06; First posted 2025-02-11 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Keratocysts of the Jaw
Keywords: Odontogenic keratocyst; topical 5-fluorouracil; modified carnoy's solution
MeSH Terms: conditions — Odontogenic Cysts | interventions — Eye Enucleation

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5-FU cream Group (Active Comparator): The entire cyst lining was radically enucleated, followed by thorough curettage of the cavity After enucleation and peripheral ostectomy a sterile radiopaque gauze coated with 5-fluorouracil cream 5% and put into the surgical cavity.
  Interventions: Procedure: Enucleation; Procedure: cyst enucleation
- Modified carnoy's solution Group (Active Comparator): The entire cyst lining was radically enucleated, followed by thorough curettage of the cavity A gauze was soaked in modified carnoy's solution and applied to the surgical cavity for 3 minutes Following the enucleation and peripheral ostectomy of the cyst.
  Interventions: Procedure: Enucleation; Procedure: cyst enucleation

INTERVENTIONS:
Procedure: Enucleation — The entire cyst lining was radically enucleated, followed by thorough curettage of the cavity with meticulous evaluation of any residual daughter cyst lining followed by reduction of lingual and buccal walls bony undercuts to remove any residual cystic epithelium
Procedure: cyst enucleation — The entire cyst lining was radically enucleated, followed by thorough curettage of the cavity with meticulous evaluation of any residual daughter cyst lining followed by reduction of lingual and buccal walls bony undercuts to remove any residual cystic epithelium.
  Using coarse round surgical carbide burs under copious normal saline irrigation, peripheral ostectomy was done for all bony walls to remove any microscopic daughter cyst, with isolation, retraction, and preservation of the lingual and inferior alveolar bundle. The bony septa were removed using rotary Lindemann fissure burs in case of multilocular lesions.
  After enucleation and peripheral ostectomy a sterile radiopaque gauze coated with 5-fluorouracil cream 5% and put into the surgical cavity.

SUMMARY:
The purpose of this study was to compare both clinically and radiographically the effect of using 5- fluorouracil cream (5-FU) versus modified carnoy's solution (MCS) as adjunctive methods in treatment of odontogenic keratocyst (OKC).

Patients and methods :This is an interventional, comparative study that was carried on 20 patients with mandibular odontogenic keratocyst and were divided randomly into two equal groups, Group I: included 10 patients in whom OKCs were treated with enucleation and peripheral ostectomy followed by application of 5-FU cream. Group II: included 10 patients in whom OKCs were treated with enucleation and peripheral ostectomy followed by application of MCS. All patients were followed up for 9 months postoperatively.

ELIGIBILITY:
Inclusion Criteria:

* patients with biopsy proved odontogenic keratocyst

Exclusion Criteria:

* relevant systemic diseases which might affect healing process.

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-10-02 (Actual); Primary Completion 2024-10-02 (Actual); Study Completion 2025-01-04 (Actual)

PRIMARY OUTCOMES:
degree of pain pain | 6 month
  degree of pain pain is measured on a visual analogue scale (VAS) started from 0 which represent (no pain at all) and end by 10 which represent (most severe pain)
swelling | 6 month
  Swelling is assessed using a vertical and horizontal references with a tape on four reference points; outer canthus of the eye, angle of the mandible, tragus, and outer corner of the mouth

SECONDARY OUTCOMES:
Quantitative computed tomography (CT) | 12 month
  Quantitative interpretation of values derived from Hounsfield units with a suitable calibration procedure is the modality of choice to determine the local bone mineral density during the follow up periods

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed K Allam, Ass prof, Principal Investigator — Tanta University
Locations (1):
- Tanta University, Tanta, Gharbia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No